CLINICAL TRIAL: NCT05145400
Title: Phase 2 Study of Isatuximab Plus Lenalidomide and Dexamethasone in Highly Toxicity-vulnerable Subjects With Newly Diagnosed Multiple Myeloma
Brief Title: Isa-Rd for Frail and/or Much Older Patients With Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1944
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Cancer
Keywords: Multiple Myeloma; isatuximab; lenalidomide; Geriatric
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — isatuximab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All subjects will receive the same treatment on the study, consisting of isatuximab, lenalidomide, and dexamethasone with 28 days cycles.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Pharmaceutical form: Solution for infusion Route of administration: Intravenous Isatuximab:10 mg/kg intravenous or 1400 mg subcutaneous (SC) via on-body delivery system (OBDS) will be administered in cycles 1-24.
Drug: Lenalidomide — Pharmaceutical form: Capsule for oral use, Route of administration: Oral Lenalidomide capsule will be given oral, the dose will be adjusted according to glomerular filtration rate (GFR): 15 mg daily if GFR > 60 mL/min, 5 mg daily if GFR 30-60 mL/min, 2.5 mg daily if GFR < 30 mL/min. Note that dialysis-dependence comprises an exclusion criterion for this study.
  Lenalidomide will be continued until disease progression, excessive toxicity or death.
  Other Names: REVLIMID
Drug: Dexamethasone — Pharmaceutical form: Tablet for oral use, Route of administration: Oral Dexamethasone tablet will be given oral: 20 mg given on days 1, 8, 15 and 22 of cycles 1-8. Administration may continue beyond cycle 8, if needed, for the prevention of infusion reactions.

SUMMARY:
This research study is investigating the safety and effectiveness of using combination of isatuximab, lenalidomide and dexamethasone for the treatment of newly diagnosed multiple myeloma (MM). The study team will use lower doses than is currently standard for these drugs. Lower doses will be used to avoid or possibly reduce any unwanted side effects commonly associated with these drugs. Using lower doses of the combination isatuximab, lenalidomide and dexamethasone, has not been approved by the Food and Drug Administration (FDA) for the treatment of newly diagnosed MM.

DETAILED DESCRIPTION:
This study aims to determine the optimal treatment regimen for older and/or otherwise toxicity-vulnerable patients with newly diagnosed multiple myeloma (NDMM) who cannot receive approved standard therapy. As a result, this Phase II trial of isatuximab, lenalidomide, and dexamethasone (Isa-Rd) selectively enroll much older and/or otherwise highly toxicity-vulnerable participants. Furthermore, the safety and effectiveness of isatuximab when used in combination with lenalidomide and dexamethasone at lower doses will be evaluated. It is expected that using this combination at lower doses, may help patients achieve a better response while causing fewer or less severe side effects.

All participants on the trial will also be evaluated by Cancer and Aging Research Group Geriatric Assessments (CARG-GA) and patient-reported outcome (PRO) measures of quality of life (QOL). "Geriatric assessment" will be referred to as "global assessment" for study purposes, to reflect the fact that younger participants will likely participate in the study. Optional correlative blood samples will be collected to study biomarkers of aging and frailty with a focus on both the relation to isatuximab specifically, as well as treatment response and risk for intolerability.

Duration of Therapy:

The length of study participation will depend on the response to the treatment, and it may last approximately 2 years. Participants will receive isatuximab for two years, and then isatuximab will be discontinued. Dexamethasone administration will occur weekly for the first eight cycles. Lenalidomide will be continued as maintenance until disease progression or unacceptable toxicity.

In the absence of treatment delays due to adverse events, treatment should continue until:

* Disease progression
* Inter-current illness that prevents further administration of treatment
* Treatment delay of more than 12 weeks.
* Unacceptable adverse event(s)
* Pregnancy
* Subject decides to withdraw from study treatment, or
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.
* Subject is lost to follow up

Duration of Follow Up:

All participants (including those withdrawn for AE (Adverse Event) will be followed after removal from study treatment until death or full subject withdrawal from the study for other reasons. Participants removed from study treatment for unacceptable AEs will be followed for resolution or stabilization of the adverse event(s).

ELIGIBILITY:
Subject Eligibility In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria

1. Written informed consent obtained to participate in the study and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information (PHI). Consent must be obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Willing and able to adhere to the study visit schedule and other protocol requirements based on the judgement of the investigator or protocol designee.
3. Predicted high risk for severe toxicity from intensive induction regimens, such as standard (full-dose) Bortezomib, cyclophosphamide, dexamethasone (VCD), lenalidomide, bortezomib, and dexamethasone (RVD), or lenalidomide and weekly dexamethasone (Rd) as each regimen was published. (Such regimens often use, for example, twice-weekly bortezomib or lenalidomide at 25 mg.) High-risk is defined as one of the following:

   1. Score ≥ 2 (indicating "frail") on the International Myeloma Working Group instrument (IMWG; Palumbo et al. [Blood 2015]),
   2. Karnofsky Performance Status (KPS) ≤ 70,
   3. Felt not to be candidate for full-intensity induction by treating clinician due to comorbidities, performance status, or other factors not otherwise captured by the Palumbo system or performance status. The reason for the subject's non-candidacy for full-intensity therapy should be described in the clinical documentation.

   Subjects qualifying for enrollment by criterion C should be discussed with the Medical Monitor before enrollment, to ensure uniform application of this criterion across participating sites.
4. Measurable MM diagnosed according to the following standard criteria. Criteria A and B must be met, in addition to C and/or D:

   1. Monoclonal plasma cells in bone marrow ≥ 10% and/or presence of biopsy-proven plasmacytoma
   2. Monoclonal protein (M-protein) present in serum and/or urine, defined as serum M-protein of ≥ 1 g/dL (0.5 g/dL for Immunoglobulin A (IgA) MM) OR urine M-protein of ≥ 200 mg/24 hours. Subjects lacking an M-protein meeting those criteria must have a serum free light chain assay with an involved light chain ≥ 10 mg/dL (100 mg/L) and an abnormal serum free light chain ratio.
   3. One or more MM-related organ dysfunction findings such as hypercalcemia, renal insufficiency, anemia, and bone lesions (CRAB) criteria listed below:

      * Calcium elevation in blood (serum calcium 1 mg/dL ≥ upper limit of normal or > 11 mg/dL)
      * Renal insufficiency (creatinine clearance < 40 ml/min or serum creatinine > 2 mg/dL)
      * Anemia (hemoglobin < 10 g/dL or ≥ 2 g/dL below normal)
      * Bone lesions (lytic bone lesions) on x-rays, computerized tomography (CT), Magnetic resonance imaging (MRI) or Positron emission tomography (PET)
   4. Myeloma-related biomarker of malignancy (1 or more should be fulfilled):

      * ≥ 60% bone marrow plasmacytosis
      * Serum involved / uninvolved free light chain ratio of ≥ 100, provided absolute level of involved light chain is at least 100 mg/L (10 mg/dL)
      * More than one focal lesion on MRI ≥ 5 mm in size
5. No prior systemic anti-myeloma therapy lasting more than 28 days (generally one cycle). Any prior therapy must be completed a minimum of 14 days before starting study drugs.
6. Subjects who require radiotherapy (which must be localized in its field size) may be treated during screening but initiating study therapy should be deferred until the radiotherapy is completed and 14 days have elapsed since the last date of radiotherapy.
7. Demonstrate adequate organ function and laboratory values as defined in below.

   Hematological
   * Hemoglobin (Hgb) ≥ 8 g/dL Transfusion of packed red blood cells or use of erythropoietin or analogs is permitted, if clinically appropriate, to achieve this threshold.
   * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L Use of growth factors is permitted to fulfill this criterion, particularly if low ANC is felt to be due to MM by treating clinician. If low ANC is felt to be due to non-MM causes, such as myelodysplasia or other bone marrow disorders unrelated to MM, then subject should not be enrolled on the study.
   * Platelets ≥ 50 × 109/L if < 50% of bone marrow nucleated cells are plasma cells, and
   * ≥ 30 × 109/L if ≥ 50% of BM (Bone Marrow) nucleated cells are plasma cells.
   * Platelet transfusions are permitted to reach entry criteria. If low platelets are felt to be due to non-MM causes, such as myelodysplasia or other bone marrow disorders unrelated to MM, then subject should not be enrolled on the study.

   Renal

   • Calculated or measured glomerular filtration rate (GFR):Any GFR as long as not currently dialysis-dependent
8. Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME (Section 5.5), at least 28 days before she starts taking lenalidomide through 30 days after the last dose of lenalidomide and 5 months after the last dose of isatuximab. FCBP must also agree to ongoing pregnancy testing during the entire duration of treatment and monthly for 5 months after the last dose of isatuximab. Men must agree to use a latex or synthetic condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 30 days after the last dose of lenalidomide and 5 months after the last dose of isatuximab. These same subjects must not donate sperm. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. All subjects enrolled into this trial, must be registered in and must comply with all requirements of the REVLIMID REMS program *A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria

1. Active infection requiring systemic antibiotics or other serious infection within 14 days prior to study treatment.
2. Subjects felt to not be candidates by treating physician for any systemic therapy due to excessive comorbidities, frailty, impaired performance status, or other severe limitations. Such limitations can be conceptualized generally as making subjects exceedingly high-risk for any systemic treatment for their MM. These limitations often stem from medical comorbidities unrelated to MM and they are hence unlikely to improve with MM therapy. The reasons for exclusion will be documented.
3. Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose excessive risk to the subject or may interfere with compliance or interpretation of the study results.
4. Light-chain (AL) amyloidosis. Subjects with secondary amyloidosis due to MM are eligible, if the amyloidosis is not felt to be a clinically significant issue (e.g., amyloid found incidentally on bone marrow core biopsy without evidence of amyloid-mediated organ compromise).
5. Myocardial infarction within 3 months prior to study treatment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
6. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
7. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study therapy that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
8. Known gastrointestinal (GI) disease that could interfere with the oral absorption or tolerance of dexamethasone or lenalidomide including difficulty swallowing.
9. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
10. Patients with a history of prior or concurrent second primary malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational treatment should generally be eligible.
11. Receiving other investigational agents less than 14 days or 5 half-lives of first dose of therapy on this protocol, whichever is longer.
12. Concurrent use of other anti-cancer agents or treatments with possible exception of agents with low likelihood of affecting outcome of this study, such as adjuvant hormonal therapy for remote history of breast cancer.
13. Known to be HIV+ or have active infection with hepatitis A, B, or C; or tuberculosis.
14. Chronic daily corticosteroids for other, non-MM-related medical conditions exceeding low-dose (e.g., prednisone ≥ 10 mg daily or equivalent).
15. Subject is receiving prohibited medications or treatments as listed in the protocol that cannot be discontinued/replaced by an alternative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From Day 1 of study treatment up to 60 months
  ORR, percentage of patients achieving a partial response or better per Revised Uniform Response Criteria by the International Myeloma Working Group (IMWG) criteria. Complete response (CR): Negative immunofixation of serum and urine, disappearance of soft tissue plasmacytomas, and <5% plasma cells in bone marrow (BM). Stringent complete response (sCR): CR plus normal free light chains (FLC) ratio and absence of clonal plasma cells in BM biopsy. Very good partial response (VGPR):-Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M component plus urine M component <100/24h. Partial response (PR) ≥50% reduction of serum M-protein & reduction in 24-hour (24h) urinary M-protein by ≥90% or to <200 mg/24h and if present at baseline, a ≥ 50% reduction in the size soft tissue plasmacytomas

SECONDARY OUTCOMES:
Treatment failure-free survival (TFFS) Time | From Day 1 of study treatment up to 60 months
  Treatment failure-free survival (TFFS): The length of time from therapy start until therapy discontinuation for any reason, including disease progression, toxicity, or death.
Progression-Free Survival (PFS) | From Day 1 of study treatment up to 60 months
  PFS is the length of time from start of study treatment until day of confirmed progression or death. The (IMWG) defines progression as any one or more: Increase of 25% from lowest response value in Serum M-protein (absolute increase (AI) ≥ 0.5 g/dL); Serum M-protein increase ≥ 1 g/dL, if lowest M component was ≥ 5 g/dL; or Urine M-protein Difference of involved & uninvolved FLC (free light chain) levels (AI > 10 mg/dL) Bone marrow plasma cell percentage irrespective of baseline status (AI ≥ 10%) New lesion(s), ≥ 50% increase from nadir, or ≥ 50% increase in longest diameter of previous lesion >1 cm in short axis; ≥ 50% increase in circulating plasma cells if only measure of disease New or definite increase in size of existing soft tissue plasmacytomas or bone lesions; Decrease in hemoglobin of ≥ 2 g/dL not related to therapy; Rise in serum creatinine by ≥2 mg/dL; Hyperviscosity related to serum paraprotein
Maximum Depth of Response | From Day 1 of study treatment up to 60 months
  Maximum depth of response (from PR to CR, including sCR) at any time will be determined based on IMWG criteria. Descriptions of partial, complete, or stringent-complete type treatment responses are summarized in the primary outcome section.
Rate of achievement of bone marrow minimal residual disease (MRD) negativity | From Day 1 of study treatment up to 60 months
  MRD status is determined by next-generation sequencing with a minimum sensitivity of 1 × 10-5. MRD refers to myeloma cells that are present in the bone marrow after a clinical response has been measured while signs and symptoms of MM are reduced or disappeared.
Clinical Benefit Rate (minimal response (MR) + ORR) | From Day 1 of study treatment up to 60 months
  The clinical benefit rate is the percentage of participants achieving overall response or minimal response. Description of overall response as defined as the percentage of subjects achieving a partial response or better (≥ PR) to study therapy at any time. Minimal response (MR) is ≥ 25% but ≤ 49% reduction of serum M-protein and reduction in 24-h urine M-protein by 50-89%. In addition to the above listed criteria, if present at baseline, a ≥ 50% reduction in the size (SPD) of soft tissue plasmacytomas is also required.
Time to Response | From Day 1 of study treatment up to 60 months
  Time to response is the length of time from start of study treatment until documentation of confirmed partial response (PR) or better based on IMWG criteria. Response description is given in the primary outcome section.
Duration of Response | From Day 1 of study treatment up to 60 months
  Duration of response is the length of time from achievement of PR or better until myeloma progression per IMWG criteria. PR description is given in the primary outcome section.
Time to Next Treatment | From Day 1 of study treatment up to 60 months
  Time to next treatment is the length of time time from start of study treatment to next MM treatment or death from any cause.
Overall Survival | From Day 1 of study treatment up to 60 months
  Overall Survival is the length of time from start of study treatment to death from any cause.
Toxicity Rate | From Day 1 of study treatment up to 60 months
  Toxicity rate is percentage of participants who experience treatment related Adverse Events (AE) as evaluated by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0. NCI-CTCAE is a descriptive terminology utilized for AE reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Tuchman, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (5):
- United States (5):
  - University of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.